CLINICAL TRIAL: NCT05134337
Title: A Phase 1, Open Label, Two-part, Fixed-sequence Drug Interaction Study to Investigate the Effect of Strong CYP3A4 Inhibitor (Itraconazole) and CYP3A4 Inducer (Rifampin) on the Pharmacokinetics of LOXO 305 in Healthy Adult Subjects
Brief Title: Study of the Effects of Itraconazole and Rifampin on LOXO-305 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20006; J2N-OX-JZNC (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-22; First posted 2021-11-24 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pirtobrutinib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (LOXO-305/Itraconazole) (Experimental): * Day 1: a single oral dose of 200 milligrams (mg) LOXO-305 was administered.
  * Day 8: oral doses of 200 mg itraconazole was administered twice daily.
  * Days 9 to 18: single oral dose of 200 mg itraconazole was administered once daily, and on Day 12 it was co-administered with a single oral dose of 200 mg LOXO-305.
  Interventions: Drug: LOXO-305; Drug: Itraconazole
- Part 2 (LOXO 305/Rifampin) (Experimental): * Day 1: a single oral dose of 200 mg LOXO-305 was administered.
  * Days 8 to 23: oral dose of 600 mg rifampin was administered once daily, and on Days 8 & 17, it was co-administered with a single oral dose of 200 mg LOXO-305.
  Interventions: Drug: LOXO-305; Drug: Rifampin

INTERVENTIONS:
Drug: LOXO-305 — Oral LOXO-305
  Other Names: Pirtobrutinib
Drug: Itraconazole — Oral itraconazole
  Arms: Part 1 (LOXO-305/Itraconazole)
Drug: Rifampin — Oral rifampin
  Arms: Part 2 (LOXO 305/Rifampin)

SUMMARY:
The main purpose of this study is to learn about how itraconazole and rifampin affect LOXO-305 in healthy participants. Participation could last about 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential.
* Within body mass index (BMI) range 18.0 to 32.0 kilograms per square meter (kg/m²).
* Participants will be in good general health, based on medical history, physical examination findings, vital signs, 12 lead electrocardiogram (ECG), or clinical laboratory tests, as determined by the Investigator (or designee).
* Able to comply with all study procedures, including the 19-night stay for those participating in Part 1 or 24-night stay for those participating in Part 2 at the Clinical Research Unit and follow-up phone call.

Exclusion Criteria:

* History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:

  * liver disease
  * pancreatitis
  * peptic ulcer disease
  * intestinal malabsorption
  * gastric reduction surgery
  * history or presence of clinically significant cardiovascular disease.
* Participants with out-of-range, at-rest vital signs.
* Abnormal laboratory values determined to be clinically significant by the Investigator (or designee).
* Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination.
* Participation in any other investigational study drug trial involving administration of any investigational drug in the past 30 days or 5 half-lives, whichever was longer, prior to the first dose administration (Day 1).
* Use or intention to use any prescription or over-the-counter medications within 14 days prior to the first dose administration (Day 1) and through end of trial.
* History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the participant at undue risk.
* Donation of blood from 56 days prior to Screening, plasma or platelets from 4 weeks prior to Screening.
* Receipt of blood products within 2 months prior to Check-in (Day -1).
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, biliary, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal (GI), neurological, or psychiatric disorder (as determined by the Investigator), or cancer within the past 5 years (except localized basal cell, squamous, or in situ cancer of the skin).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renée Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2 (LOXO 305/Rifampin): * Day 1: a single oral dose of 200 mg LOXO-305 was administered
  * Days 8 to 23: oral dose of 600 mg rifampin was administered once daily, and on Days 8 & 17, it was co-administered with a single oral dose of 200 mg LOXO-305.
Period: Overall Study
Arm/Group | Part 1 (LOXO-305/Itraconazole) | Part 2 (LOXO 305/Rifampin)
Started | 15 | 12
Received at Least One Dose of Study Drug | 15 (3 participants discontinued the study after receiving the LOXO-305 dose on Day 1. Therefore, the safety analysis population for the Itraconazole alone and the LOXO-305 + Itraconazole treatment sequences includes only the remaining 12 participants.) | 12
Completed | 12 | 12
Not Completed | 3 | 0
Not completed — Subject Discontinued Out of Precaution Due to Covid-19 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (LOXO-305/Itraconazole) | Part 2 (LOXO 305/Rifampin) | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (9.13) | 40.9 (7.79) | 39.2 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of LOXO-305
Description: Cmax of LOXO-305
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on days 1 and 12
Population: All part 1 participants who received a dose of LOXO-305 on day 1, itraconazole with LOXO-305 on day 12, had at least one quantifiable plasma concentration of LOXO-305, and had at least one PK parameter computed for the specified timepoints. Participants were excluded from the analysis if they experienced an AE of vomiting that occurred at or before 2 times the median time to maximum observed plasma concentration (Tmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 (LOXO-305/Itraconazole)
Number analyzed (Participants) | 15
nanogram per milliliter (ng/mL)
  Day 1 | 4000 (23.5)
  Day 12: number analyzed (Participants) | 12
  Day 12 | 4100 (17.2)

2. Primary Outcome: Part 1: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of LOXO 305
Description: PK: AUC0-t of LOXO 305
Time Frame: as for outcome 1
Population: All part 1 participants who received a dose of LOXO-305 on day 1, itraconazole with LOXO-305 on day 12, had at least one quantifiable plasma concentration of LOXO-305, and had at least one PK parameter computed for the specified timepoints. Participants were excluded from the analysis if they experienced an AE of vomiting that occurred at or before 2 times the median Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 (LOXO-305/Itraconazole)
Number analyzed (Participants) | 15
hour*nanogram per milliliter (h*ng/mL)
  Day 1 | 80000 (23.4)
  Day 12: number analyzed (Participants) | 12
  Day 12 | 122000 (22.7)

3. Primary Outcome: Part 1: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of LOXO-305
Description: AUC0-inf of LOXO-305
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 (LOXO-305/Itraconazole)
Number analyzed (Participants) | 15
hour*nanogram per milliliter (h*ng/mL)
  Day 1 | 80800 (23.4)
  Day 12: number analyzed (Participants) | 12
  Day 12 | 123000 (23.4)

4. Primary Outcome: Part 2: PK: Maximum Observed Plasma Concentration (Cmax) of LOXO-305
Description: Cmax of LOXO-305
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on days 1 and 17; Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose on day 8
Population: All part 2 participants who received a dose of LOXO-305 on day 1, rifampin with LOXO-305 on day 8 and day 17, had at least one quantifiable plasma concentration of LOXO-305, and had at least one PK parameter computed for the specified timepoints. Participants were excluded from the analysis if they experienced an AE of vomiting that occurred at or before 2 times the median Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 2 (LOXO 305/Rifampin)
Number analyzed (Participants) | 12
nanogram per milliliter (ng/mL)
  Day 1 | 4480 (20.4)
  Day 8 | 4170 (15.6)
  Day 17 | 2580 (22.4)

5. Primary Outcome: Part 2: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of LOXO 305
Description: PK: AUC0-t of LOXO 305
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 2 (LOXO 305/Rifampin)
Number analyzed (Participants) | 12
hour*nanogram per milliliter (h*ng/mL)
  Day 1 | 79700 (17.6)
  Day 8 | 48500 (14.7)
  Day 17 | 23000 (20.1)

6. Primary Outcome: Part 2: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of LOXO-305
Description: AUC0-inf of LOXO-305
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on days 1 and 17
Population: All part 2 participants who received a dose of LOXO-305 on day 1, rifampin with LOXO-305 on day 17, had at least one quantifiable plasma concentration of LOXO-305, and had at least one PK parameter computed for the specified timepoints. Participants were excluded from the analysis if they experienced an AE of vomiting that occurred at or before 2 times the median Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 2 (LOXO 305/Rifampin)
Number analyzed (Participants) | 12
hour*nanogram per milliliter (h*ng/mL)
  Day 1 | 80600 (17.3)
  Day 17 | 23600 (19.8)

7. Primary Outcome: Part 2: PK: Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours Postdose (AUC0-24) of LOXO-305
Description: AUC0-24 of LOXO-305
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose on days 1 and 8
Population: All part 2 participants who received a dose of LOXO-305 on day 1, rifampin with LOXO-305 on day 8, had at least one quantifiable plasma concentration of LOXO-305, and had at least one PK parameter computed for the specified timepoints. Participants were excluded from the analysis if they experienced an AE of vomiting that occurred at or before 2 times the median Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 2 (LOXO 305/Rifampin)
Number analyzed (Participants) | 12
hour*nanogram per milliliter (h*ng/mL)
  Day 1 | 50200 (14.5)
  Day 8 | 48600 (14.7)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (up to day 28 for Part 1; up to day 33 for Part 2)
Description: All participants who received at least 1 dose of study drug. The adverse events were analyzed and reported according to the treatment sequences pre-specified in the statistical analysis plan (SAP).
Groups:
- Part 1: 200 mg LOXO-305 Alone; Part 2: 200 mg LOXO-305 Alone: Participants with adverse events observed during or after Day 1 LOXO-305 dosing and prior to Day 8 dosing were grouped under this arm.
- Part 1: 200 mg Itraconazole Alone: Participants with adverse events observed during or after Day 8 itraconazole dosing and prior to Day 12 dosing were grouped under this arm.
- Part 1: 200 mg LOXO-305 + 200 mg Itraconazole: Participants with adverse events observed during or after Day 12 LOXO-305 and itraconazole dosing were grouped under this arm.
- Part 2: 200 mg LOXO-305 (Day 8) + 600 mg Rifampin: Participants with adverse events observed during or after Day 8 LOXO-305 and rifampin dosing and prior to Day 17 dosing were grouped under this arm.
- Part 2: 200 mg LOXO-305 (Day 17) + 600 mg Rifampin: Participants with adverse events observed during or after Day 17 LOXO-305 and rifampin dosing were grouped under this arm.
Arm/Group | Part 1: 200 mg LOXO-305 Alone | Part 1: 200 mg Itraconazole Alone | Part 1: 200 mg LOXO-305 + 200 mg Itraconazole | Part 2: 200 mg LOXO-305 Alone | Part 2: 200 mg LOXO-305 (Day 8) + 600 mg Rifampin | Part 2: 200 mg LOXO-305 (Day 17) + 600 mg Rifampin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 2/12 | 1/12 | 0/12 | 0/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: 200 mg LOXO-305 Alone (N=15) | Part 1: 200 mg Itraconazole Alone (N=12) | Part 1: 200 mg LOXO-305 + 200 mg Itraconazole (N=12) | Part 2: 200 mg LOXO-305 Alone (N=12) | Part 2: 200 mg LOXO-305 (Day 8) + 600 mg Rifampin (N=12) | Part 2: 200 mg LOXO-305 (Day 17) + 600 mg Rifampin (N=12)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT05134337/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT05134337/SAP_001.pdf